CLINICAL TRIAL: NCT05243615
Title: Internet-delivered Cognitive Behavioural Therapy for Persons With Stroke: Randomized Controlled Trial
Brief Title: Internet-delivered Cognitive Behavioural Therapy for Persons With Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Swati Mehta, Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12132
Record Dates: First submitted 2022-02-07; First posted 2022-02-17 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Stroke; Depression; Anxiety
Keywords: Stroke; Depression; Anxiety; internet-delivered cognitive behaviour therapy
MeSH Terms: conditions — Stroke; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke internet delivered cognitive behavioural therapy (Experimental): A 10-week internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants who have sustained a stroke. In addition to the online program, a Guide with experience delivering ICBT will provide support by email or phone call once a week. The Guide will spend approximately 15 minutes per week/per client.
  Interventions: Behavioral: Guided internet delivered cognitive behavioural therapy
- Stroke Rehabilitation Education (Active Comparator): A 10-week stroke-specific rehabilitation education program for stroke patients in usual care at specialized stroke rehabilitation units. The lessons will include information on spinal cord injury rehabilitation: 1)stroke basics, 2)mental health after stroke, 3)pain after stroke, 4)understanding rehabilitation 5)summary of lessons through an online platform. A Guide will check in with participants once a week to answer any content-related questions. The Guide will spend approximately 15 minutes per week/per client.
  Interventions: Behavioral: Stroke rehabilitation mental health education

INTERVENTIONS:
Behavioral: Guided internet delivered cognitive behavioural therapy — A 10-week internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants who have sustained a stroke. In addition to the online program, a Guide with experience delivering ICBT will provide support by email or phone call once a week. The Guide will spend approximately 15 minutes per week/per client.
  Arms: Stroke internet delivered cognitive behavioural therapy
Behavioral: Stroke rehabilitation mental health education — A 10-week stroke-specific rehabilitation education program for stroke patients in usual care at specialized stroke rehabilitation units. The lessons will include information on spinal cord injury rehabilitation: 1)stroke basics, 2)mental health after stroke, 3)pain after stroke, 4)understanding rehabilitation 5)summary of lessons through an online platform. A Guide will check in with participants once a week to answer any content-related questions. The Guide will spend approximately 15 minutes per week/per client.
  Arms: Stroke Rehabilitation Education

SUMMARY:
Approximately 30% of people with stroke experience symptoms of depression. Many may benefit from access to mental health services that target unhelpful thoughts, such as cognitive behaviour therapy (CBT), but go untreated due to lack of access to specialized care, costs, remote location, or stigma related to seeking care. Internet Cognitive Behavioural Therapy (ICBT) may overcome these barriers. The stroke ICBT program teaches skills such as challenging unhelpful thoughts, memory and attention, managing related physical symptoms, and pacing through a mix of online learning and weekly contact with a trained Guide. While the program's content was found to be acceptable among individuals after stroke, the program's effectiveness still needs to be evaluated. Thus, the primary purpose of this study is to evaluate if the stroke ICBT program will improve symptoms of depression compared to an attention control group. Individuals in both groups will answer questions about themselves and their injury and describe symptoms of depression, quality of life, and health service use to evaluate its impact on people's wellbeing. The study results will be useful in determining if the ICBT program is effective and whether it should be part of routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* Canadian residents;
* diagnosed with a stroke at least 6 months ago;
* endorsing symptoms of depression (PHQ-9≥5); 5) suicide risk score <8 (Suicide Behaviours Questionnaire);
* speak and read English;
* able to access and be comfortable using computers and the internet;
* willing to provide a physician as an emergency contact.

Exclusion Criteria:

* significant cognitive impairment, a score of <21 on the Telephone Interview for Cognitive Status;
* aphasia, with significant language impairment;
* currently involved in another psychotherapeutic intervention;
* present with a severe mental health disorder requiring in-person therapy (e.g., severe suicidal ideation, severe substance abuse, a recent history of psychosis or mania).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Change in depression | baseline, 10 weeks, 3 months
  Measured by Patient Health Questionnaire - 9 Item (PHQ-9), higher scores indicate worse outcomes
Change in anxiety | baseline, 10 weeks, 3 months
  Measured by Generalize Anxiety Disorder - 7 Item (GAD7)higher scores indicate worse outcomes

SECONDARY OUTCOMES:
Change in quality of life symptoms | baseline, 10 weeks, 3 months
  Measured by VAS on the EuroQol-5D (EQ5D), higher scores indicate better outcomes
Self-efficacy | baseline, 10 weeks, 3 months
  Measured by Self-Efficacy for managing Chronic Disease-6 (SEMCD), higher scores indicate better outcomes
Change in perceived disability | baseline, 10 weeks, 3 months
  Measured by The World Health Organization Disability Assessment Schedule ,(WHODAS), higher scores indicate worse outcomes
Treatment credibility | baseline, 10 weeks
  Measured by Treatment Credibility Questionnaire (TCQ) which contains 4 items. The first three items range from 0-9 with higher scores indicating better outcome, and the fourth item ranges from 0-100%, with higher scores indicating greater improvement in functioning.
Treatment satisfaction | baseline, 10 weeks
  Measured by Internet-CBT Treatment Satisfaction Measure, higher scores indicate greater satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Robert Teasell, MD, Principal Investigator — Western University

IPD SHARING:
Plan to Share IPD: No